CLINICAL TRIAL: NCT05122871
Title: Scape Room With High Fidelity Simulator: Results in the Learning and Satisfaction of Nursing Degree Students
Brief Title: Scape Room With High Fidelity Simulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Cristina Franco Antonio, Associate Professor of nursing studies, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16/2021
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Nursing Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scape room (Experimental)
  Interventions: Other: Scape Room
- Simulation (Active Comparator)
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Scape Room — Practical training through scape-room with simulator
  Arms: Scape room
Other: Simulation — Practical training through simulator
  Arms: Simulation

SUMMARY:
The objective of the present study is assess the efficcacy in the acquisition of knowledge and practical skills of a scape room with high definition simulators.

An experimental trial will be carried out in which the students of the intervention group will receive practical training on newborn care in the delivery room through the development of a scape room with high-fidelity simulators. The control group students will receive practical training only with the use of high-fidelity simulators. The participants of both groups will previously receive a theoretical training of 10 hours. Knowledge acquisition and student satisfaction with both methodologies will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Nursing degree students of University of Extremadura

Exclusion Criteria:

* 1st year nursing degree students
* Nursing degree students of other universities

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge test | 1 month after training session
  The degree of knowledge and skills related to the care of the newborn will be measured by means of an evaluation questionnaire that will consist of 20 multiple choice questions..

SECONDARY OUTCOMES:
Satisfaction likert scale | 1 month after training session
  the degree of student satisfaction with the methodology used will be evaluated with a 6-item likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Franco Antonio, PhD, Principal Investigator — University of Extremadura
Locations (1):
- Cristina Franco Antonio, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No